CLINICAL TRIAL: NCT02294435
Title: Visceral Manifold and Unitary Device Study for the Repair of Thoracoabdominal Aortic Aneurysms
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sanford Health (Other)
Collaborators: Dakota Vascular (Other)
Responsible Party: Principal Investigator, Patrick Kelly, Vascular Surgeon, Dakota Vascular
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SH VMS
Record Dates: First submitted 2014-11-14; First posted 2014-11-19 (Estimated); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Thoracoabdominal Aneurysms
Keywords: Thoracoabdominal Aneurysms; Endovascular; Ps-ide; Early Feasibility; Aneurysm; Aortic Aneurysm, Thoracic; Aortic Aneurysm; Aortic Diseases; Cardiovascular Diseases; Vascular Diseases; Pararenal aneurysm; Juxtarenal aneurysm; Aortic dissection; Short neck infrarenal aneurysm; Type 4 thoracoabdominal; TAAA
MeSH Terms: conditions — Aneurysm; Aortic Aneurysm, Thoracic; Aortic Aneurysm; Aortic Diseases; Cardiovascular Diseases; Vascular Diseases; Aortic Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Primary Study Arm (Experimental): The TAAA Debranching Stent Graft System is comprised of two investigational devices including the Thoracic Bifurcation and the Visceral Manifold and the Unitary Manifold. The thoracic bifurcation and the visceral manifold as well as the unitary manifold work to facilitate endovascular stenting of the visceral vessels (renals, celiac, SMA) while maintaining flow to the visceral and infrarenal segments.
  Interventions: Device: Visceral Manifold and Thoracic Bifurcation; Device: Unitary Manifold
- Expanded Selection Arm (Experimental): The expanded selection arm is for subjects not eligible for open repair or other endovascular options due to comorbidities or anatomical limitations and do not meet inclusion in the primary study arm. The Thoracic Bifurcation and the Visceral Manifold as well as the Unitary Manifold work to facilitate endovascular stenting of the visceral vessels (renals, celiac, SMA) while maintaining flow to the visceral and infrarenal segments.
  Interventions: Device: Visceral Manifold and Thoracic Bifurcation; Device: Unitary Manifold

INTERVENTIONS:
Device: Visceral Manifold and Thoracic Bifurcation — Visceral Manifold and Thoracic Bifurcation Endovascular stent graft system
Device: Unitary Manifold — Unitary Manifold Endovascular stent graft system

SUMMARY:
The primary objective of the Visceral Manifold and Unitary Device Study is to assess the use of the thoracic bifurcation and the visceral manifold or the unitary device to repair thoracoabdominal aortic aneurysms in patients having appropriate anatomy. The primary intent of the study is to assess safety and preliminary effectiveness of the device. Additionally, the study will assess technical success and treatment success at each follow-up interval.

DETAILED DESCRIPTION:
The primary objective of the clinical investigation Visceral Manifold and Unitary Device Study is to assess the use of the thoracic bifurcation and the visceral manifold or the unitary stent graft system to repair thoracoabdominal aortic aneurysms in patients having appropriate anatomy. The primary intent of the study is to assess safety (i.e. freedom from major adverse events (MAE) at 30 days) and preliminary effectiveness (i.e., treatment success and technical success) of the device (i.e., the proportion of treatment group subjects that achieve and maintain treatment success at one year). Additionally, the study will assess technical success and treatment success at each follow-up interval.

ELIGIBILITY:
Inclusion Criteria:

* An aneurysm with a maximum diameter of ≥ 5.5 cm or 2 times the normal diameter just proximal to the aneurysm using orthogonal (i.e., perpendicular to the centerline) measurements
* Aneurysm with a history of growth ≥ 0.5 cm in 6 months
* Saccular aneurysm deemed at significant risk for rupture
* Symptomatic aneurysm greater than or equal to 4.5 cm
* Axillary or brachial and iliac or femoral access vessel morphology that is compatible with vascular access techniques, devices or accessories, with or without use of a surgical conduit
* Proximal landing zone for the thoracic bifurcation stent graft:

  •≥ 2.5 cm of nonaneurysmal aortic segment including previously placed graft material (neck) distal to the left subclavian artery (LSA)
  * Diameter in the range of 26-42 mm
  * Adequate distance from the celiac artery, in order to accommodate cannulation from the antegrade access point when considering the total deployed length of the thoracic bifurcation and visceral manifold
* Proximal landing zone for the unitary manifold stent graft:

  * Nonaneurysmal aortic segment including previously placed graft material (neck) with a minimum seal zone length of 3 cm
  * Diameter in the range of 19-32 mm
* Iliac artery or aortic distal fixation site greater than or equal to 15 mm in length and diameter in the range of 8 - 25 mm
* Age: ≥ 18 years old
* Life expectancy: > 1 year

Exclusion Criteria:

General exclusion

* Patient is a good candidate for and elects for open surgical repair
* Can be treated in accordance with the instructions for use with a legally marketed
* Is eligible for enrollment in a manufacturer-sponsored IDE at the investigational site
* Unwilling to comply with the follow-up schedule
* Inability or refusal to give informed consent
* Urgent or emergent presentation
* Patient is pregnant or breastfeeding
* Patient has a contained rupture
* Patient has a ruptured aneurysm
* Patient has a dissection in the portion of the aorta intended to be treated
* Obstructive stenting of any or all of the visceral vessels
* Poor performance status including two major system failures (cardiovascular, pulmonary, renal, hepatobiliary, and neuromuscular)

Medical exclusion criteria

* Known sensitivities or allergies to the materials of construction of the devices, including nitinol (Nickel:Titanium), polyester, platinum-iridium, polytetrafluoroethylene (PTFE)
* Known hypersensitivity or contraindication to anticoagulation or contrast media that cannot be adequately medically managed
* Uncorrectable coagulopathy
* Body habitus that would inhibit x-ray visualization of the aorta or exceeds the safe capacity of the equipment
* Patient has had a major surgical or interventional procedure unrelated to the treatment of the aneurysm planned < 30 days of the endovascular repair
* Unstable angina (defined as angina with a progressive increase in symptoms, new onset at rest or nocturnal angina)
* Systemic or local infection that may increase the risk of endovascular graft infection
* Baseline creatinine greater than 2.0 mg/dL
* History of connective tissue disorders (e.g., Marfan Syndrome, Ehler's Danlos Syndrome)
* Prior aneurysm repair that would involve relining of the previously placed graft material requiring placement of the investigational system in a landing zone that expands beyond any limits of the previously placed graft material

Anatomical exclusion criteria

* Minimum branch vessel diameter less than 5 mm
* Thrombus or excessive calcification within the neck of the aneurysm
* Anatomy that would not allow maintenance of at least one patent hypogastric artery
* Anatomy that would not allow primary or assisted patency of the left subclavian artery

Expanded Selection Arm Inclusion Criteria

Patient that meets the criteria for inclusion in the primary study arm but has one or more of the following criteria which would exclude them from the primary study arm:

* Minimum branch vessel diameter less than 5 mm
* Urgent or emergent presentation
* Patient has a contained rupture
* Patient has a ruptured aneurysm
* Patient has a type B dissection (subacute or chronic) in the portion of the aorta intended to be treated
* Poor performance status including two major system failures (cardiovascular, pulmonary, renal, hepatobiliary, and neuromuscular)
* Baseline creatinine greater than or equal to 2.0 mg/dL
* Anatomy that would not allow for maintenance of at least one hypogastric artery
* Anatomy that would not allow for primary or assisted patency of the left subclavian artery
* Prior aneurysm repair that would involve relining of the previously placed graft material requiring placement of the investigational system in the a landing zone that expands beyond any limits of the previously placed graft material
* Obstructive stenting of any or all of the visceral vessels

OR

Patient that meets criteria for inclusion in the primary study arm and:

* Would not be eligible for the primary study arm per a documented reason other than those outlined above, and
* Per the opinion of the Principal Investigator, with concurrence of the IRB, alternative therapies are unsatisfactory and the probable risk of using the investigational device is no greater than the probable risk from the disease or condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2015-02 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Freedom from major adverse events (MAEs) at 30 days | 30 days
  Major adverse events include death, bowel ischemia, myocardial infarction, paraplegia, renal failure, respiratory failure, and stroke.

SECONDARY OUTCOMES:
Treatment success and technical success at 1 year | 1 year
  Treatment success is defined as a composite of technical success and freedom from the following:
  * Aneurysm enlargement
  * Aneurysm rupture
  * Aneurysm-related mortality
  * Conversion to open repair
  * Secondary intervention for migration, Type I and III endoleaks, device integrity failure , and patency-related events
Treatment success at various timepoints | 1 month, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  Treatment success and the individual components of treatment success including freedom from the following:
  * Aneurysm enlargement
  * Aneurysm-related mortality
  * Aneurysm rupture
  * Conversion to open repair
  * Secondary intervention for migration, type I and III endoleaks, device integrity failure, and patency-related events.
  * Renal failure
  * All-cause mortality
  * Endoleaks
  * Device integrity failure
  * Patency-related events
  * Other device-related events

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Kelly, MD, Principal Investigator
Locations (1):
- Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson J, Nykamp M, Danielson L, Remund T, Kelly PW. A novel endovascular debranching technique using physician-assembled endografts for repair of thoracoabdominal aneurysms. J Vasc Surg. 2014 Nov;60(5):1177-1184. doi: 10.1016/j.jvs.2014.05.090. Epub 2014 Jul 3. PMID 24997805
- [Derived] Jorgensen BD, Malek M, VandenHull A, Remund T, Truong KC, Pohlson K, Kelly PW. A novel physician-assembled endograft for the repair of pararenal, paravisceral, Crawford type IV thoracoabdominal aortic aneurysms, and aneurysms requiring treatment after prior repair. J Vasc Surg. 2020 Dec;72(6):1897-1905.e2. doi: 10.1016/j.jvs.2020.03.045. Epub 2020 Apr 23. PMID 32335306